CLINICAL TRIAL: NCT05523895
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Pimavanserin for the Treatment of Irritability Associated With Autism Spectrum Disorder
Brief Title: Pimavanserin for the Treatment of Irritability Associated With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-069
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Irritability Associated With Autism Spectrum Disorder
Keywords: Randomized; Placebo-controlled
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo given once daily, as one capsule matching in size and color the respective pimavanserin treatment
  Interventions: Drug: Placebo
- Pimavanserin low dose (Experimental): Patients aged 5 to 12 years: 10 mg/day pimavanserin Patients aged 13 to 17 years: 20 mg/day pimavanserin
  Pimavanserin given once daily, as capsule of 10 or 20 mg dose strength, respectively, according to the patient's age
  Interventions: Drug: Pimavanserin
- Pimavanserin high dose (Experimental): Patients aged 5 to 12 years: 20 mg/day pimavanserin Patients aged 13 to 17 years: 34 mg/day pimavanserin
  Pimavanserin given once daily, as capsule of 20 or 34 mg dose strength, respectively, according to the patient's age
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin
  Other Names: Nuplazid
  Arms: Pimavanserin high dose; Pimavanserin low dose
Drug: Placebo — Pimavanserin matching placebo
  Arms: Placebo

SUMMARY:
6-week, randomized, double-blind, fixed-dose, placebo-controlled, parallel group study in children and adolescents (aged 5 to17 years) with autism spectrum disorder (ASD) with irritability, agitation, or self-injurious behaviors to study the efficacy and safety of pimavanserin

DETAILED DESCRIPTION:
This study will be conducted as a 6-week, randomized, double-blind, fixed-dose, placebo-controlled, parallel group study in children and adolescents (5 through 17 years of age) with ASD with irritability, agitation, or self-injurious behaviors.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female and 5 through 17 years of age
* Informed consent prior to the conduct of any study procedures
* Patients (to the best of his/her ability), parent/legally accepted representative, and designated caregiver (if applicable) are able to understand the nature of the study, follow protocol requirements, and be willing to comply with study drug administration requirements
* Able to swallow a test placebo capsule without difficulty
* Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ASD (APA 2013) and diagnosis is confirmed by the Autism Diagnostic Interview-Revised (ADI-R)
* Score ≥18 on the Irritability subscale of the Aberrant Behavior Checklist (ABC)
* Score ≥4 (moderate or greater severity) on the Clinical Global Impression-Severity (CGI-S) of irritability score
* No current comorbid psychiatric disorder other than attention-deficit hyperactivity disorder (ADHD) or anxiety disorder
* Drug-naïve to antipsychotic treatment (or <2 weeks antipsychotic treatment for any reason), or prior lack of tolerability to adequate dose of any duration of antipsychotic confirmed by caregiver and medical records review
* If patient is undergoing concurrent behavioral therapy for autism related symptoms or behaviors, this non-pharmacological treatment regimen has been stable for at least 4 weeks, and will be consistent throughout the study
* For female patients only: unable to become pregnant or agree to use a highly effective non-hormonal method of contraception. Females of childbearing potential must have a negative pregnancy test

EXCLUSION CRITERIA:

* Requires treatment with a medication prohibited by the protocol, including concomitant psychotropic drugs targeting irritability, including those used off-label (clonidine, guanfacine, and propranolol; lithium, valproate), medications that prolong the QT interval, and strong cytochrome P450 (CYP) 3A4 enzyme (CYP3A4) inhibitors and inducers
* Changes in medications or medication doses (for medical and allowed comorbid psychiatric conditions) in the last 4 weeks
* Any known history of angioedema, serotonin or neuroleptic malignant syndromes, dystonic reaction, or tardive dyskinesia, due to an antipsychotic or psychotropic medication
* At a significant risk of suicide, or is a danger to self or others
* At risk of significant violent behavior to the extent that participation would pose an undue risk to other patients, caregivers, or others
* Positive urine drug test
* Met DSM-5 criteria for substance use disorders within the last 6 months
* Confirmed genetic disorder associated with ASD, a cognitive and/ or behavioral disturbance or profound intellectual disability (IQ ≤50)
* History of seizures, unless seizure-free and off epileptic drugs for at least 6 months
* Any condition that, in the opinion of the Investigator, would interfere with the ability to comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk
* Current evidence, or history within the last 12 weeks, of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies
* Weight <15 kg
* History or presence on at least one ECG of protocol-defined cardiac conduction abnormalities
* Known family or personal history or symptoms of long QT syndrome or history of cardiac arrhythmias or risk factors for torsade de pointes and/or sudden death, including symptomatic bradycardia, hypokalemia or hypomagnesemia, and presence of congenital prolongation of the QT interval
* Any member of the household has suffered from COVID-19 or had a COVID-19 (PCR or immunoglobulin) positive test in the last 4 weeks
* One or more clinical laboratory test value outside of protocol-defined limits
* Breastfeeding or lactating, or has a positive pregnancy test result (for patients of childbearing potential)
* Sensitivity to pimavanserin or any of the excipients
* Participating in another clinical study of any investigational drug, device, or intervention
* Participated in greater than 2 interventional pharmaceutical clinical research studies in the last 6 months
* Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (18):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Cortica Inc. (Glendale), Glendale, California
  - Cortica Inc. (San Rafael), San Rafael, California
  - 1st Allergy and Clinical Research Group, d/b/a IMUNOe Research Centers, Centennial, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - The EHS Medical Practice, PA, D/B/A Sarkis Clinical Trials, Gainesville, Florida
  - APG Research, LLC, Orlando, Florida
  - AMR Baber Research Incorporated, Naperville, Illinois
  - Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada
  - ERG Clinical Research - New York, PLLC DBA Richmond Behavioral Associates, Staten Island, New York
  - Quest Therapeutics of Avon Lake dba Haidar Almhana Nieding LLC, Avon Lake, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Relaro Medical Trials, LLC, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - AIM Trials, LLC, Plano, Texas
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington
- Australia (3):
  - Children's Health Queensland Hospital and Health Service, South Brisbane, QDL
  - Monash Health, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- France (4):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Centre de Ressources Autisme Rhône-Alpes - Center Hospitalier le Vinatier, Bron
  - CHU de Nantes, Nantes
  - L'Assistance Publique - Hôpitaux de Paris, labélisé Institut Carnot, Paris
- Hungary (4):
  - Vadaskert Hospital, Budapest
  - Magyarországi Református Egyház Bethesda Gyermekkórháza, Budapest
  - Békés Megyei Központi Kórház, Gyula
  - Szegedi Tudományegyetem, Szeged
- Italy (11):
  - Azienda Ospedaliero Universitaria (AOU) Consorziale Policlinico, Bari
  - La Nostra Famiglia - Scientifica IRCCS Eugenio Medea, Bosisio Parini
  - The Childhood and Adolescence Neuropsychiatry Clinic - University of Cagliari and Pediatric Hospital "A. Cao" - ASL 8 of Cagliari, Cagliari
  - Policlinico Riuniti - Azienda Ospedaliero Universitaria, Foggia
  - IRCCS Istituto Giannina Gaslini, Genova
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino - IRCCS, Pavia
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Azienda Ospedaliera-Universitaria Senese, Siena
  - Azienda Ospedaliera Universitaria Integrata di Verona (AOUI), Verona
- Poland (6):
  - Gdańskie Centrum Zdrowia Sp. z o.o., Gdansk
  - Centrum Badań Klinicznych PI-House Sp. z o.o., Gdansk
  - NAVICULA - Centrum Diagnozy i Terapii Autyzmu, Lodz
  - Ginemedica Sp. Zoo, S.K., Wroclaw
  - Centrum Neuropsychiatrii NEUROMED SP ZOZ, Wroclaw
  - MedicMental Indywidualna Specjalistyczna Praktyka Lekarska Monika Szewczuk-Boguslawska, Wroclaw
- Serbia (4):
  - Institute of Mental Health, Belgrade
  - University Clinical Center Kragujevac, Clinic for Psychiatry, Kragujevac
  - University Clinical Center Nis, Center for Mental Health, Niš
  - Clinical Center of Vojvodina, Clinic for Psychiatry, Novi Sad
- Spain (7):
  - Hospital General de Alicante, Alicante
  - Institut Global d´Atenció Integral del Neurodesenvolupament (IGAIN), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Complejo Asistencial Universitario de Burgos, Burgos
  - Hospital Universitario Infanta Leonor, Madrid
  - Complejo Asistencial de Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Pimavanserin-matching placebo, given as 1 capsule once daily
- Pimavanserin Low Dose: Pimavanserin given as 1 capsule once daily. Patients aged 5-12 years: 10 mg/day; patients aged 13-17 years: 20 mg/day
- Pimavanserin High Dose: Pimavanserin given as 1 capsule once daily. Patients aged 5-12 years: 20 mg/day; patients aged 13-17 years: 34mg/day
Period: Overall Study
Arm/Group | Placebo | Pimavanserin Low Dose | Pimavanserin High Dose
Started | 78 | 78 | 81
Completed | 74 | 67 | 75
Not Completed | 4 | 11 | 6
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Noncompliance with study drug | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Not further specified | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All patients randomised
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin Low Dose | Pimavanserin High Dose | Total
Number analyzed (Participants) | 78 | 78 | 81 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.88) | 9.8 (3.54) | 9.8 (3.11) | 9.8 (3.18)
Age, Customized [Count of Participants; unit: Participants]
  5-12 years | 63 | 61 | 64 | 188
  13-17 years | 15 | 17 | 17 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 13 | 53
  Male | 57 | 59 | 68 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 5 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 8 | 12 | 11 | 31
  White | 61 | 56 | 58 | 175
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Hungary | 6 | 7 | 5 | 18
  United States | 39 | 38 | 40 | 117
  Poland | 18 | 19 | 21 | 58
  Italy | 2 | 3 | 5 | 10
  France | 6 | 1 | 4 | 11
  Australia | 4 | 1 | 2 | 7
  Serbia | 3 | 5 | 3 | 11
  Spain | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 6 in Caregiver-rated Aberrant Behavior Checklist Irritability (ABC-I) Subscale Score
Description: The Aberrant Behavior Checklist (ABC) is a caregiver-rated scale comprised of 5 empirically-derived subscales encompassing 58 items that describe various behavior problems. It measures domains of irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech. ABC-I is one of the subscales and comprises of 15 items. Minimum score is 0, maximum is 45. A score for each item ranges from 0 indicating "not at all a problem" to 3 indicating "the problem is severe in degree". Subscale scores are calculated by summing the items within that subscale. Higher scores indicate greater impairment.
Time Frame: 6 weeks
Population: Full Analysis Set: all randomized patients who received at least one dose of study drug and have a baseline value and at least one post-baseline value for the ABC-I subscale score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pimavanserin Low Dose | Pimavanserin High Dose
Number analyzed (Participants) | 72 | 64 | 74
score on a scale | -9.6 (1.06) | -11.2 (1.09) | -11.2 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Pimavanserin Low Dose; Test type: Superiority; p = 0.2986, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-4.6 to 1.4], Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: Placebo vs Pimavanserin High Dose; Test type: Superiority; p = 0.2859, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-4.5 to 1.3], Standard Error of Mean 1.49

ADVERSE EVENTS:
Time Frame: From screening to end of safety follow-up, which was to be performed at 10 weeks, i.e. 4 weeks after last dose of study drug
Arm/Group | Placebo | Pimavanserin Low Dose | Pimavanserin High Dose
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/77 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/77 | 0/81
Other Adverse Events (participants affected / at risk) | 11/78 | 17/77 | 16/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | Pimavanserin Low Dose (N=77) | Pimavanserin High Dose (N=81)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | Pimavanserin Low Dose (N=77) | Pimavanserin High Dose (N=81)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (7) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 5 (6)
Somnolence (Nervous system disorders) | 4 (4) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05523895/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT05523895/SAP_001.pdf